CLINICAL TRIAL: NCT01376336
Title: Randomized Controlled Trial of Safe Water Storage Among People Living With HIV
Brief Title: Trial of Safe Water Storage Among People Living With HIV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: University of Zambia (Other)
Responsible Party: Joe Brown/Lecturer, London School of Hygiene and Tropical Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: QA308
Record Dates: First submitted 2011-06-14; First posted 2011-06-20 (Estimated); Last update posted 2011-06-20 (Estimated); Status verified 2011-06

CONDITIONS: Diarrhea; Waterborne Disease; HIV
Keywords: environmental health; diarrhea; water; HIV
MeSH Terms: conditions — Diarrhea; Waterborne Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Safe storage device (Experimental): This arm will be assigned a safe water storage device.
  Interventions: Device: Safe storage device
- Control (No Intervention): This arm of the trial will receive nothing until the end of the trial.

INTERVENTIONS:
Device: Safe storage device — This device is a specially designed water storage container that is intended to reduce the likelihood of re-contamination of household stored drinking water.
  Arms: Safe storage device

SUMMARY:
Environmental health-related pathogens include faecal-oral, diarrhoeagenic microbes that may be transmitted via drinking water and are related to sanitation and hygiene. Previous research has suggested that safeguarding household drinking water against recontamination may be a critical intervention that can reduce risks of diarrheal diseases and may be especially important for people living with HIV/AIDS (PLWHA) and other vulnerable populations (Clasen et al. 2007). The investigators propose here a randomised, controlled trial of a household safe storage container for drinking water in a well defined, HIV-impacted population in peri-urban Lusaka, Zambia. After a baseline data collection period (9 months) half of all households (150 households) will be given a safe water storage container specifically designed to prevent recontamination of water in household use. All households will be followed for an additional 9 months. Results of this study will help determine whether this promising water quality intervention can reduce diarrhoea and related outcomes in this and similar vulnerable populations.

DETAILED DESCRIPTION:
Specific Aim #1: To assess environmental health-related risk and outcomes in a low income peri-urban area of Zambia with a high percentage of people living with HIV/AIDS (PLWHA) (longitudinal observational cohort study and baseline) (Year 1). We will assemble a rich dataset on environmental health-related risk factors in a well defined population, with a focus on household drinking water quality and other water, sanitation, and hygiene (WSH) exposures.

Specific Aim #2: To quantify the WSH-related disease burden among PLWHA, compared with those without HIV/AIDS (individual and household level stratification) (conclusion of baseline). After nine months of data collection, we will perform an initial analysis to determine WSH-related risk by HIV status.

Specific Aim #3: To assess the impact of a water quality intervention on the longitudinal prevalence of Highly Credible Gastrointestinal Illness (HCGI) among PLWHA (randomized controlled trial, year 2). We will conduct a randomised, controlled trial of a safe water storage intervention. We will assess the health impacts of this intervention, with particular focus on the high-risk groups of PLWHA and children under 5 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Resident of Misisi compound, Lusaka
* Willing to participate in the study
* Is able to give informed consent and does so
* Household has one or more children who are aged 48 months or less at the start of the trial
* The household stores drinking water in the home

Exclusion Criteria:

* Not a resident of Misisi compound, Lusaka
* Unwilling to participate in the study
* Unable to give informed consent or chooses not to participate
* Household does not have one or more children aged 48 months or less at the start of the trial
* The household does not store drinking water in the home

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1600 (Estimated)
Dates: Start 2011-08; Primary Completion 2013-08 (Estimated); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
Self-reported diarrheal disease | 18 months
  Self-reported diarrheal disease information will be collected from each study participant monthly. These data will be collected monthly with 24 hour, 48 hour, and 7-day recall. Data will be assessed at 18 months (change from baseline).

SECONDARY OUTCOMES:
Weight-for-age z-score | 18 months
  Weight-for-age z-scores will be taken for all children who are aged less than 48 months ("under 5s") at the start of the trial and monthly during the trial. These data are useful in tracking short-term wasting, associated with diarrheal disease events. Data will be assessed at 18 months (change from baseline).
E. coli and total coliforms in household drinking water | 18 months
  Microbiological indicators of fecal contamination of drinking water at the household level. Samples will be taken from all households monthly. Data will be assessed at 18 months (change from baseline).
Salivary antibody response | 18 months
  We will collect salivary samples from all consenting individuals (an additional consent form is required) to gather information on IgG and IgA response to specific diarrheal pathogens using a multiplex assay. This measure provides useful information on both outcomes of interest (diarrheal disease) and exposure to diarrheagenic pathogens. Samples will be taken at three time points: the beginning, midpoint, and end of the trial. Data will be assessed at 18 months (change from baseline).

CONTACTS AND LOCATIONS:
Overall Officials: Joe Brown, PhD, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (1):
- Tropical Gastroenterology and Nutrition Group (TROPGAN), University of Zambia School of Medicine, Lusaka, Zambia